CLINICAL TRIAL: NCT02200445
Title: A Phase I Study of Low Dose Subcutaneous Interleukin-2 (IL-2) For The Treatment of Ulcerative Colitis.
Brief Title: Low Dose IL-2 for Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scott B. Snapper, MD PHD (Other)
Responsible Party: Sponsor-Investigator, Scott B. Snapper, MD PHD, Associate Professor of Medicine, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00009599; 2015P000016 (Other: Brigham & Women's Hospital, Boston MA)
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Results first posted 2020-12-19 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2022-08

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Inflammatory bowel disease; Interleukin 2; Interleukin-2; IL-2; Regulatory T Cells; Tregs; T-Lymphocytes, Regulatory
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interleukin-2 (Experimental): Study drug: Interleukin-2 (aldesleukin, Proleukin, IL-2).
  Each subject will receive an 8-week course of once-daily, subcutaneously administered IL-2. There will be three dose cohorts. Each subject will be recruited into a single dose cohort and receive a single dose level of IL-2 throughout the study.
  The dose levels will be as follows:
  * Cohort 1: 0.3x10^6 IU/m^2/day.
  * Cohort 2: 1.0x10^6 IU/m^2/day.
  * Cohort 3: 1.5x10^6 IU/m^2/day.
  Up to 6 subjects will be recruited to each dose cohort.
  Once the maximum effective dose has been identified, a further 10 subjects will receive IL-2 at the maximum effective dose.
  Interventions: Drug: Interleukin-2 (aldesleukin).

INTERVENTIONS:
Drug: Interleukin-2 (aldesleukin). — Description of intervention is covered in "Arm", above.
  Other Names: Proleukin.

SUMMARY:
The purpose of this study is to determine the safety and maximum effective dose (MED) of Interleukin-2 in subjects with moderate-to-severe ulcerative colitis.

DETAILED DESCRIPTION:
Interleukin-2 (IL-2) is a T cell growth factor. IL-2 is currently licensed for the treatment of metastatic renal cell carcinoma and metastatic melanoma, where it promotes the expansion of anti-cancer cytotoxic T cells and natural killer (NK) cells. However at low doses (100-times lower than those used in cancer therapy), IL-2 promotes the selective expansion of regulatory T cells (Tregs): an immune modulating subset of CD4+ lymphocytes.

A recent phase 1 clinical trial from our collaborators at the Dana Farber Cancer Institute showed that low-dose IL-2 selectively expands Tregs in patients with treatment-resistant Graft vs. Host Disease (GvHD), and that low-dose IL-2 is safe in this condition. A detailed immunological analysis of samples from this study showed that low-dose IL-2 treatment was associated with increased Treg proliferation, increased de novo thymic generation of Tregs, and a resolution of defects in intracellular signalling and apoptosis seen in Tregs in chronic GvHD. A recent phase 1 study from another group showed that low-dose IL-2 is safe in the treatment of HCV-associated vasculitis. Low-dose IL-2 has also been shown to be well-tolerated in subjects with HIV.

Ulcerative colitis (UC) is a chronic inflammatory disease of the colon. Evidence from pre-clinical models of intestinal inflammation, and also from patients with monogenetic defects in Treg function, suggests that Tregs play a role in the prevention of inflammation in the intestine.

The treatment (or intervention) in this study is a once-daily, subcutaneous injection of IL-2, for a total of 8 weeks. The first 2 doses of the study drug will be administered by research nurses at Boston Children's Hospital. Further doses will be self-administered, at home. Training will be provided for correct self-administration.

This is a 3+3 dose escalation study of IL-2 in moderate-to-severe UC. This study design is powered to identify the MED of low-dose IL-2 in UC. Once the MED is identified, a further 10 subjects will receive IL-2 at that dose. Recruitment of between 2 and 28 patients is planned. The maximum tolerated dose (MED) is the highest tolerated dose level at which a minimum of 6 subjects have been evaluated, with fewer than 2 evaluable subjects in 6 experiencing a dose limiting toxicity (DLT); i.e. DLT in >1/6 evaluable subjects. In addition to the above at least 1 patient should meet the criteria for response or remission for it to be considered the MED.

Dose levels are based on the experience of our collaborators in GvHD. In addition to determining the MED, this study will determine if low-dose IL-2 is safe and well-tolerated in patients with moderate-to-severe ulcerative colitis. A detailed immunological analysis of samples obtained from this study will determine if low-dose IL-2 expands Tregs in vivo, in patients with moderate-to-severe UC. Immunological changes will then be correlated with clinical response.

The study will take place at Boston Children's Hospital. The study will involve 10 study visits. Most of the study visits involve blood tests. A flexible sigmoidoscopy or colonoscopy will be performed as part of the screening process. A flexible sigmoidoscopy will also be performed on completion of therapy, to determine clinical response.

The first two subjects to receive the study drug will be admitted overnight following the first dose. Subsequent doses will be administered on an out-patient basis. All other subjects will receive IL-2 on an out-patient basis.

Responders (with an acceptable side-effect profile) will be allowed to continue the study drug for at least 1 year. Compensation will be provided for participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years.
* A diagnosis of UC made by standard clinical, radiological, endoscopic and histological criteria.
* Moderate to severe UC with a Mayo score of 6-12.
* Failure to tolerate or failure to respond to at least one conventional therapy with the intention of inducing or maintaining remission (examples include oral corticosteroids, oral 5-aminosalicylates, azathioprine and/or 6-mercaptopurine, or a tumor necrosis factor (TNF) antagonist). Corticosteroid dependency (inability to taper oral corticosteroids without a recurrence of disease activity) is also included in this category.
* Stable doses of concomitant medications.
* A negative pregnancy test in the 2 weeks prior to anticipated commencement of the study drug, in female subjects of child-bearing age. Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.
* Ability to provide informed consent.

Exclusion Criteria:

* A diagnosis of Crohn's disease or Inflammatory Bowel Disease - Unspecified (IBD-U, a diagnostic classification formerly termed "indeterminate colitis").
* Requirement for immediate surgical, endoscopic or radiological intervention for toxic megacolon, massive hemorrhage, perforation, sepsis, or intra-abdominal or perianal abscess.
* Ileostomy, proctocolectomy or subtotal colectomy with ileorectal anastomosis.
* History of colorectal cancer or dysplasia.
* Positive stool test for Clostridium difficile.
* Current medically significant infection.
* Significant laboratory abnormalities, including;

  1. Hb < 8.0 g/dL, WBC < 2.5 x 103/mm3, Plt < 100 x 103/mm3.
  2. Creatinine ≥ 1.5x institutional upper limit of normal (ULN).
  3. Total bilirubin > 2.0 mg/dL, ALT > 2x institutional ULN, GGT > 2x institutional ULN. Elevated unconjugated bilirubin related to Gilbert's syndrome is allowed.
  4. Abnormal thyroid function tests.
* Positive serology for HIV, hepatitis B virus (HBV) or HCV.
* Positive screening test for tuberculosis (TB).
* First dose of an anti-TNF medication within 4 weeks of anticipated study commencement, or a subsequent dose within 2 weeks of commencement; or ciclosporin or tacrolimus within 2 weeks of anticipated study commencement.
* Received another investigational new drug (IND) within 5 half-lives of that agent before the planned commencement of SC IL-2.
* Malignancy within the last 5 years.
* Allergy to any component of the study drug.
* Pregnant or lactating women.
* Inability to comply with the study protocol or inability to give informed consent.
* Prior exposure to IL-2.
* Uncontrolled cardiac angina or symptomatic congestive cardiac failure (NYHA Class III or IV).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-02; Primary Completion 2020-10-01 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Snapper, MD PhD, Principal Investigator — Boston Children's Hospital; Jessica R Allegretti, MD, MPH, Study Director — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koreth J, Matsuoka K, Kim HT, McDonough SM, Bindra B, Alyea EP 3rd, Armand P, Cutler C, Ho VT, Treister NS, Bienfang DC, Prasad S, Tzachanis D, Joyce RM, Avigan DE, Antin JH, Ritz J, Soiffer RJ. Interleukin-2 and regulatory T cells in graft-versus-host disease. N Engl J Med. 2011 Dec 1;365(22):2055-66. doi: 10.1056/NEJMoa1108188. PMID 22129252
- [Background] Matsuoka K, Koreth J, Kim HT, Bascug G, McDonough S, Kawano Y, Murase K, Cutler C, Ho VT, Alyea EP, Armand P, Blazar BR, Antin JH, Soiffer RJ, Ritz J. Low-dose interleukin-2 therapy restores regulatory T cell homeostasis in patients with chronic graft-versus-host disease. Sci Transl Med. 2013 Apr 3;5(179):179ra43. doi: 10.1126/scitranslmed.3005265. PMID 23552371
- [Background] Saadoun D, Rosenzwajg M, Joly F, Six A, Carrat F, Thibault V, Sene D, Cacoub P, Klatzmann D. Regulatory T-cell responses to low-dose interleukin-2 in HCV-induced vasculitis. N Engl J Med. 2011 Dec 1;365(22):2067-77. doi: 10.1056/NEJMoa1105143. PMID 22129253
- [Background] Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med. 1987 Dec 24;317(26):1625-9. doi: 10.1056/NEJM198712243172603. PMID 3317057
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095

RESULTS

PARTICIPANT FLOW:
Groups:
- Interleukin-2 Dose A: Study drug: Interleukin-2 (aldesleukin, Proleukin, IL-2).
  The dose levels will be as follows:
  * Cohort 1: 0.3x10^6 IU/m^2/day.
- Interleukin-2 Dose B: - Cohort 2: 1.0x10^6 IU/m^2/day.
- Interleukin-2 Dose C: - Cohort 3: 1.5x10^6 IU/m^2/day
Period: Overall Study
Arm/Group | Interleukin-2 Dose A | Interleukin-2 Dose B | Interleukin-2 Dose C
Started | 4 | 17 | 5
Completed | 3 | 13 | 3
Not Completed | 1 | 4 | 2
Not completed — Lack of Efficacy | 1 | 2 | 2
Not completed — Adverse Event | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interleukin-2 Dose A | Interleukin-2 Dose B | Interleukin-2 Dose C | Total
Number analyzed (Participants) | 4 | 17 | 5 | 26
Age, Continuous [Mean (Full Range); unit: years] | 36.7 [27 to 57] | 43 [18 to 69] | 46.6 [25 to 71] | 38.7 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 1 | 8
  Male | 2 | 12 | 4 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 16 | 5 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 17 | 5 | 26
Extent [Count of Participants; unit: Participants]
  Ulcerative Proctitis | 1 | 1 | 0 | 2
  Left-sided | 2 | 12 | 3 | 17
  Pancolitis | 1 | 4 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious and Non-serious Adverse Events.
Description: Enumeration of the serious and non-serious adverse events seen in the study. Enumeration of any dose limiting toxicity seen in the study.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Interleukin-2 Dose A | Interleukin-2 Dose B | Interleukin-2 Dose C
Number analyzed (Participants) | 4 | 17 | 5
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Clinical Response
Description: A decrease from baseline in the total Mayo score of at least 3 points and at least 30% , with an accompanying decrease in the subscore for rectal bleeding of at least 1 point or an absolute subscore for rectal bleeding of 0 or 1
Time Frame: 8 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Interleukin-2 Dose A | Interleukin-2 Dose B | Interleukin-2 Dose C
Number analyzed (Participants) | 4 | 17 | 5
Participants
  Clinical response criteria met | 1 | 9 | 0
  Clinical Response criteria not met | 2 | 5 | 3
  withdrew from trial | 1 | 3 | 2

3. Secondary Outcome: Number of Participants With Clinical Remission
Description: A total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Interleukin-2 Dose A | Interleukin-2 Dose B | Interleukin-2 Dose C
Number analyzed (Participants) | 4 | 17 | 5
Participants
  Clinical Remission criteria met | 0 | 4 | 0
  Clinical Remission criteria not met | 3 | 9 | 3
  withdrew from trial | 1 | 4 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline of study until subjects withdrew, were lost to follow-up, or completed the study up to week 8 and through the OLE up to week 52.
Arm/Group | Interleukin-2 Dose A | Interleukin-2 Dose B | Interleukin-2 Dose C
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/17 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/17 | 0/5
Other Adverse Events (participants affected / at risk) | 4/4 | 17/17 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interleukin-2 Dose A (N=4) | Interleukin-2 Dose B (N=17) | Interleukin-2 Dose C (N=5)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 3 (6) | 9 (9) | 5 (6)
Papular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
achiness/chills (General disorders) | 0 (0) | 3 (3) | 2 (2)
joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Flushing (General disorders) | 0 (0) | 1 (1) | 0 (0)
macular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
pityriasis rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczematous rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
numbness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrush (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1) | 0 (0)
fever (General disorders) | 0 (0) | 8 (8) | 4 (4)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1) | 0
migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
IBD Flare (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Increased Bowel Movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
strep throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT02200445/Prot_SAP_000.pdf